CLINICAL TRIAL: NCT07147335
Title: The Role of Serum AKR1B10 in Early Warning of Hepatocellular Carcinoma in Cirrhosis Patients ------ Risk Early Warning and Follow-up Study
Brief Title: The Role of Serum AKR1B10 in Early Warning of Hepatocellular Carcinoma in Cirrhosis Patients
Acronym: AKR1B10
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Principal Investigator, Zhongtian Peng, Executive Director, The First Affiliated Hospital of University of South China
Other Study IDs: AKR1B10's clinical study
Record Dates: First submitted 2025-08-12; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis; Hepotacellular Carcinoma
Keywords: AKR1B10; Hepotacellular carcinoma; cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Biospecimen Description: blood (2 mL) was collected in a plain VACUTAINER tube containing no anticoagulant and allowed to clot at room temperature for 30 minutes, followed by centrifugation at 1,500g for 10 minutes at 4°C to remove clots. Supernatants (serum) were immediately transferred into clean polypropylene tubes (200 µL per tube) using a Pasteur pipette, encoded with a number, and stored or transported at -80°C. Serum samples that were hemolyzed, icteric, or lipemic were excluded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The serum AKR1B10 concentration was high in patients with cirrhosis.: The serum AKR1B10 concentration was high in patients with cirrhosis.
  Interventions: Diagnostic Test: serum AKR1B10 levels
- The serum AKR1B10 concentration was low in patients with cirrhosis: The serum AKR1B10 concentration was low in patients with cirrhosis
  Interventions: Diagnostic Test: serum AKR1B10 levels

INTERVENTIONS:
Diagnostic Test: serum AKR1B10 levels — Investigators collected blood from the patients every three months to test their serum AKR1B10 levels.

SUMMARY:
Hepatocellular carcinoma (HCC) is a globally prevalent malignancy. In its characteristic "chronic hepatitis-liver cirrhosis-HCC" progression trilogy, patients with cirrhosis demonstrate a 5-year HCC incidence rate of 3%-5%, yet effective monitoring strategies remain lacking. Current early diagnosis relies on the combination of imaging techniques and serum alpha-fetoprotein (AFP), but AFP measurements are frequently confounded by pregnancy and liver diseases, resulting in suboptimal sensitivity and specificity. In recent years, novel tumor biomarkers such as AKR1B10 (Aldo-keto reductase family 1 member B10) have been examined. This multicenter prospective cohort study aims to validate the predictive value of serum AKR1B10 for malignant transformation in cirrhosis-HCC progression, and evaluate its combined efficacy with existing risk prediction models, ultimately establishing a high-sensitivity early diagnostic strategy for clinical implementation.

DETAILED DESCRIPTION:
Patients with liver cirrhosis and chronic hepatitis were enrolled in this clinical trial. The study was designed to investigate the clinical value of serum AKR1B10 in hepatocellular carcinoma (HCC) risk prediction, early diagnosis, and screening among individuals with cirrhosis. Previous studies have demonstrated elevated AKR1B10 levels in small tumor nodules measuring <2 cm. Based on these findings, Investigators hypothesize that in a subset of cirrhotic patients, hepatic tissues may harbor ultra-early carcinogenic or precancerous lesions undetectable by current clinical modalities, and that serum AKR1B10 could serve as an early warning signal for such occult malignant transformation.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for liver cirrhosis and chronic hepatitis
* Aged 18-75 years, regardless of gender
* Willing to participate in the study and provides signed informed consent
* Has not participated in other clinical trials within the last 3 months

Exclusion Criteria:

* Pregnancy or lactation
* Incomplete clinical data, serological or imaging records
* Lost to follow-up prior to reaching the observational endpoints
* Aged <18 years or >75 years
* Concurrent severe systemic diseases (e.g., involving cardiovascular, cerebral, pulmonary, renal, or hematopoietic systems)
* Current or recent (within 3 months) participation in other clinical trials
* Diagnosed with hepatocellular carcinoma (HCC)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Hepatitis and Liver Cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
HCC | 36 mouths
  In this clinical trial, all patients with cirrhosis underwent ultrasound and serum AKR1B10 tests every three months

CONTACTS AND LOCATIONS:
Locations (1):
- University of South China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeo YH, Lee YT, Tseng HR, Zhu Y, You S, Agopian VG, Yang JD. Alpha-fetoprotein: Past, present, and future. Hepatol Commun. 2024 Apr 12;8(5):e0422. doi: 10.1097/HC9.0000000000000422. eCollection 2024 May 1. PMID 38619448
- [Background] Cao W, Chen HD, Yu YW, Li N, Chen WQ. Changing profiles of cancer burden worldwide and in China: a secondary analysis of the global cancer statistics 2020. Chin Med J (Engl). 2021 Mar 17;134(7):783-791. doi: 10.1097/CM9.0000000000001474. PMID 33734139
- [Background] Ilikhan SU, Bilici M, Sahin H, Akca AS, Can M, Oz II, Guven B, Buyukuysal MC, Ustundag Y. Assessment of the correlation between serum prolidase and alpha-fetoprotein levels in patients with hepatocellular carcinoma. World J Gastroenterol. 2015 Jun 14;21(22):6999-7007. doi: 10.3748/wjg.v21.i22.6999. PMID 26078578
- [Background] Allemani C, Matsuda T, Di Carlo V, Harewood R, Matz M, Niksic M, Bonaventure A, Valkov M, Johnson CJ, Esteve J, Ogunbiyi OJ, Azevedo E Silva G, Chen WQ, Eser S, Engholm G, Stiller CA, Monnereau A, Woods RR, Visser O, Lim GH, Aitken J, Weir HK, Coleman MP; CONCORD Working Group. Global surveillance of trends in cancer survival 2000-14 (CONCORD-3): analysis of individual records for 37 513 025 patients diagnosed with one of 18 cancers from 322 population-based registries in 71 countries. Lancet. 2018 Mar 17;391(10125):1023-1075. doi: 10.1016/S0140-6736(17)33326-3. Epub 2018 Jan 31. PMID 29395269
- [Background] Kapoor S. AKR1B10 and its emerging role in tumor carcinogenesis and as a cancer biomarker. Int J Cancer. 2013 Jan 15;132(2):495. doi: 10.1002/ijc.27685. Epub 2012 Jul 30. No abstract available. PMID 22729709
- [Background] Ye X, Li C, Zu X, Lin M, Liu Q, Liu J, Xu G, Chen Z, Xu Y, Liu L, Luo D, Cao Z, Shi G, Feng Z, Deng H, Liao Q, Cai C, Liao DF, Wang J, Jin J, Cao D. A Large-Scale Multicenter Study Validates Aldo-Keto Reductase Family 1 Member B10 as a Prevalent Serum Marker for Detection of Hepatocellular Carcinoma. Hepatology. 2019 Jun;69(6):2489-2501. doi: 10.1002/hep.30519. Epub 2019 Apr 6. PMID 30672601
- [Background] Chidambaranathan-Reghupaty S, Fisher PB, Sarkar D. Hepatocellular carcinoma (HCC): Epidemiology, etiology and molecular classification. Adv Cancer Res. 2021;149:1-61. doi: 10.1016/bs.acr.2020.10.001. Epub 2020 Nov 28. PMID 33579421
- [Background] Zhu AX. Hepatocellular carcinoma: are we making progress? Cancer Invest. 2003 Jun;21(3):418-28. doi: 10.1081/cnv-120018233. PMID 12901288